CLINICAL TRIAL: NCT02949102
Title: Effects of Gymnemic Acids Lozenge on Reward Region Response to Receipt and Anticipated Receipt of High-Sugar Food, High-Sugar Food Pictures, and Ad Lib Candy Intake
Brief Title: Crave Crush Neuroimaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: Cravecrush (Unknown); Oregon Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FOUR002
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crave Crush (Experimental): Crave Crush is a plant-based tablet that alters taste perception by affecting sweet taste receptors on the tongue.
  Interventions: Dietary Supplement: Crave Crush
- Placebo (Placebo Comparator): The placebo tablet is comparable in taste and is comprised primarily of sorbitol.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Crave Crush — Crave Crush is a dietary supplement that affects sweet taste receptors on the tongue.
  Arms: Crave Crush
Dietary Supplement: Placebo — The placebo tablet is comparable in taste and is comprised primarily of sorbitol.
  Arms: Placebo

SUMMARY:
The purpose of the research is to test whether a gymnemic acids (GA) lozenge will reduce reward region response to intake of high-sugar food and ad lib candy intake and whether the GA lozenge reduced reward region response to anticipated intake of high-sugar food and high-sugar food pictures relative to a placebo lozenge.

DETAILED DESCRIPTION:
Test the hypothesis that an acute dose of Crave Crush will produce greater reductions in reward region response to a taste of a high-sugar/high-fat beverage and anticipated receipt of this beverage than a placebo dose.

Test the hypothesis that a dose of Crave Crush will result in reduced ad lib candy intake while the participants complete a survey after the fMRI scan. Participants will receive a second dose of Crave Crush or placebo. They will then be placed in a room to complete a few surveys. A bowl of candy will be placed on the table. Participants will be told that the candy is left over from their assessment and that they are free to have as much as they like, because the candy must be discarded after each participant.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years old
* report having a sweet tooth
* report desire to lose weight
* Body Mass Index between 18 and 40

Exclusion Criteria:

* major psychiatric disorders
* serious health problems (e.g., diabetes)
* habitual use of psychoactive drugs or medications
* contraindications for MRI scanning (e.g., ferromagnetic braces)
* gluten or lactose intolerance
* a vegan diet.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
fMRI responses to high-sugar food tastes and food cues | 13 minutes
  Blood oxygen dependent signal (BOLD) response in exposure to intake of high-sugar food and food cues will be measured during a fMRI scan to test whether the GA lozenge produces greater reductions in activity in reward-related brain regions relative to a placebo lozenge.

SECONDARY OUTCOMES:
candy consumption | 15 minutes
  The current study tested whether the GA lozenge reduces ad lib candy intake relative to a placebo lozenge.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, Ph.D., Principal Investigator — Oregon Research Behavioral Intervention Strategies

IPD SHARING:
Plan to Share IPD: No